# **Study title:**

Efficacy of Emotionally Focused Therapy Among Spanish Speaking Couples [E(f)FECTS]

# **Unique Protocol ID:**

E(f)FECTS

## **NCT ID:**

Not yet assigned

## **Document:**

Informed Consent Form for Study Participants (English and Spanish versions)

**Ethics Committee Approval:** 

November 11, 2021

## **Informed Consent Form for Study Participants – ENGLISH VERSION**

**TITLE OF RESEARCH STUDY**: Emotionally Focused Therapy for Couples: A Clinical Trial in Spanish Speaking countries

STUDY INVESTIGATORS: Martiño Rodríguez-Gonzalez, Ph. D.<sup>1</sup>, Jonathan Sandberg, Ph.D.<sup>2</sup>, Alfonso Osorio, Ph.D. <sup>1</sup>, Shayne Anderson, Ph.D.<sup>2</sup>, Paul Greenman, Ph.D.<sup>3</sup>, Marie-France Lafontaine Ph.D.<sup>4</sup>, Patrick Steffen, Ph.D.<sup>2</sup>, María Calatrava, Ph.D. <sup>1</sup>, María del Pilar Martínez-Díaz Ph.D. <sup>5</sup> and graduate students from UNAV or BYU, [<sup>1</sup>University of Navarra (UNAV), <sup>2</sup>Brigham Young University (BYU), <sup>3</sup>University of Québec au Outaouais (UQO), <sup>4</sup>University of Ottawa (UO), <sup>5</sup>Comillas Pontifical University]

Dr. Martiño Rodríguez-Gonzalez (Ph.D.), who is a marriage and family therapist and full-time researcher at the Institute for Culture and Society (ICS) at the University of Navarra, is the primary supervisor for this research study. Dr. Rodríguez-Gonzalez can be reached by mail at: Edificio de Bibliotecas. E-31009. Universidad de Navarra. Pamplona (Spain) and by phone at: +34 948 425600 Ext. 802367, or by email at: effects@unav.es

| Participant Name: _ |
|---------------------|
| Date: |

#### INTRODUCTION

You are being asked to take part in a research study. Before you decide to be part of this research study, you need to understand the risks and benefits of participation so that you can make an informed decision. This is known as informed consent. This consent form will give you information about the research study and what your participation will involve. If you would like more information about something mentioned here, or if you have any other questions, please feel free to ask (Dr. Rodríguez-Gonzalez, who can be reached by mail at: Edificio de Bibliotecas. E-31009. Universidad de Navarra. Pamplona. Spain. Phone at: +34 948 425600 Ext. 802367, or by e-mail at: effects@unav.es).

Once you understand what the research study involves, you will be asked to sign this consent form if you still desire to take part in this research study. You are free to choose whether or not to take part in the research study. Also, you are free to withdraw from this research study at any time, even after the study has begun. If you withdraw, as a couple you will be reimbursed \$100 for each stage of the study completed during your participation (\$50 to each member of the couple; from this it will be necessary to subtract the costs in case of an international transaction and/or currency exchange). Since we are examining how couples change over the process of therapy, if you choose not to participate in the research components of this study (e.g., questionnaires), you will not be assigned a therapist nor provided complementary couples therapy; however, we will provide you with a list of available community services in your area should you desire.

Before you sign this form, please ask questions on any aspects of this research study that are unclear to you. You may take as much time as necessary to think this over.

#### PURPOSE OF THIS RESEARCH STUDY

This research study is designed to develop a better understanding of how Spanish speaking individuals in Spanish speaking countries are impacted through the process of couple therapy. The purpose of the research study is to assess whether a particular therapy model, the Emotionally Focused Therapy, can help Spanish speaking couples develop a closer relationship with their partner and to learn how to maintain this closeness after therapy is completed.

#### **PROCEDURE**

Research Participation: What does participation in the study entail?

During this visit, if you decide to sign the consent form and participate in the study, you will be asked to complete a series of questionnaires and a personal interview with one of the investigators/therapists of the study, to confirm you understand what your participation will entail and to clarify and determine final eligibility requirements (some information may be difficult to accurately assess through online questionnaires and/or over a phone/video call). In these questionnaires you will be asked about your personality, moods, health, and yourself as well as about your relationship with your partner. This personal interview will require about 30-40 minutes (15-20 minutes per partner separately).

If after the first visit you are still eligible to participate in the therapy study, you will be notified of your eligibility via e-mail and/or a phone call within 2-5 business days. If you are not deemed eligible, you will not be included in the study, but you will be provided with a list of community resources for couple therapy in your area. Regardless of your eligibility, your scores (comprised of your responses to the initial evaluation assessments) will be kept for future comparisons in the study with other participants/potential participants. All identifying information will be removed from your responses to ensure anonymity and confidentiality.

Once deemed eligible, you will be randomly be assigned, with your partner, to either a control group or a treatment group. If assigned to the control group, you will be asked to complete a series of periodic assessments as well as to participate in a follow-up phase with one or more member(s) of the research team through occasional phone calls over a 5- to 7-month period. At the end of this process you will be offered, along with your partner, the opportunity to participate in a complementary psycho-educational weekend program for couples. This program is also based on the Emotionally Focused Therapy model and is called the "hold me tight" workshop.

If you are assigned to the treatment group, you will be asked to participate in 20 sessions of couples therapy each 75 minutes in length. These sessions will take place on a weekly basis (with some possible exceptions). As part of your participation in the study, before and/or after said therapy sessions, you will be asked to complete a series of questionnaires that are part of the elements of the project associated with this research. All therapy sessions will occur at a couple therapy clinic in your area.

Regardless of assignment to the treatment group or the control group, each set of questionnaires should take no more than 10 minutes to complete. In some cases, instead of a paper-pencil questionnaire, participants will be requested to respond online (in the therapy setting or at home).

## Couple Therapy

If you are placed in the treatment group, you will be assigned to an experienced therapist from your area who will call you to arrange your first therapy appointment together with your partner. You will be seen for a total of 20 sessions that will each last approximately 1 hour and 15 minutes each. You and your partner will be required to attend therapy together each week, except at some point between sessions 2 and 5, where your assigned therapist will hold an individual session with you and a separate session with your partner. Sessions will be conducted by therapists trained in Emotionally Focused Therapy (EFT). Supervision of the therapy process will be carried out by approved supervisors of EFT. All sessions will be videotaped and/or audio-taped for supervision and research purposes.

Your decision to participate in this study, implies that you agree to the research framework of the study as well, which entails agreeing to video recordings of all therapy sessions, and completing the questionnaires which are given to you. As a participant, you are free to end your participation in the study at any point. However, so long as you have agreed to participate and are still participating in the study, you acknowledge that you do so having a familiarity of the nature of the study.

## Therapeutic Approach Used in This Research Study

The specific approach of couples counseling that you will be offered is called Emotionally Focused Therapy for Couples. Emotionally Focused Therapy for Couples views relationship distress as resulting from negative patterns of interaction that couples develop over time. Emotionally Focused Therapy helps couples step out of negative patterns so that they can help each other establish safety and connection within their relationship. It also teaches partners' how to better request and respond to one another's needs for support and love. Scientific research studies have consistently demonstrated that this form of therapy is very helpful in helping distressed couples improve their relationships, and that these improvements last long after therapy has been completed.

## What will it cost me to participate? Will I be paid for participating?

There will be <u>no</u> cost associated with participation in any part of this research study. As a couple, you will be paid \$60.00 per hour of participation (payment is for participation in the research portion of the study, not for attending therapy sessions), with an estimated total of 7 hours of participation in the research portion depending on the group to which you are assigned. If this participation requires more than 7 hours, you will be paid, as a couple, \$80 for each additional hour.

Finally, those couples assigned to the treatment group will be asked to participate in a final follow-up phase once the therapeutic interventions have been completed (the 20 therapy sessions). This follow up will not be required for couples in the control group, who will participate in the psychoeducational intervention based on the EFT model (called "hold me tight"). Follow-up assessments will take place at 3, 6, 12, 18 and 24 months after the therapeutic intervention has been completed. Participating couples who complete the first two follow-up assessments, which will take place at 3 and 6 months, will receive \$70 (per couple), an additional \$70 for completing the 12- and 18-month assessment, and a final \$70 for completing the 24-month assessment after the end of the therapy.

## **RISKS AND BENEFITS**

## **Risks**

Therapy involves answering questions about thoughts and emotions, as does the completion of study questionnaires. Participants might experience some mild discomfort in responding to them, but no more so than if they were to remember a sad event in their lives. If for any reason this were to happen and the discomfort were to become difficult to manage, participants who are receiving EFT will be encouraged to discuss this difficulty with their therapist, who will be a qualified mental health professional. Participants in the control group will be given the contact information for Dr. Martiño Rodríguez-González, who is a registered psychologist, should they wish to address any discomfort that might arise.

## Benefits

The benefits of participating in EFT are well-established. These include improvement in one's relationship with their partner as well as one's mood and overall psychological state.

## **CONFIDENTIALITY**

All information collected as a result of this study will be treated in such a way as to maximize confidentiality and protection of your personal information. Completed questionnaires, counsellors' progress notes, and the audio and/or video records used in this study will be kept in a locked filing cabinet at the psychotherapy clinic/site at which your therapy sessions are held¹. All online questionnaires will be completed and stored on a secure and encrypted server. Furthermore, this information will be sent to the University of Navarra through a secure and encoded communications channel. No names or personal information linking your identity to your responses or your partner's will be placed on the questionnaires nor the video records. Your names will be known only to the personnel who are directly involved in the research study. These include the study investigators, the clinical supervisors, and your therapist. Anonymity will be assured through the pooling of all data so that the published results will be presented in group format and no individual or couple will be identified.

<sup>&</sup>lt;sup>1</sup> The paper-pencil questionnaires must be kept at the psychotherapy clinic/site of the therapists in charge of the process with every couple, in a locked filing cabinet.

In some situations, however, a member of the research team must break this confidentiality agreement<sup>2</sup>. These exceptions are in cases of a court order, of imminent danger to yourself or to others, of disclosures of child abuse, or of disclosures of abuse by a health care professional. In terms of child abuse, we are required by law to inform the appropriate authorities if we become aware that any child under the age of 18 is being abused or at risk of being abused. So, while this does not relate to any disclosures of your own childhood abuse experiences, it would be necessary for us to file a report with the proper authorities if you disclose that your abuser was still in regular, unsupervised contact with young children.

## Data storage for research purposes

The digital copy of the paper-pencil questionnaires (that you will answer in in your therapist's office) and the list linking couple identification numbers and names, as well as other contact information (e.g., e-mail), will be kept in a hard-disk with password in a separate locked filing cabinet in Dr. Rodríguez-González's office for a period of 5 years after the completion of the study, at which point they will be destroyed. Only the principal investigator, Dr. Rodríguez-González, will have access to this information.

All other printed and electronic files (not mentioned in the previous paragraph) related to this research project (e. g., data matrix with the questionnaires codified or videotaped therapy sessions) will be kept in a hard-disk with password in a separate locked filing cabinet in Dr. Rodríguez-González's office (UNAV) for a period of 15 years (2035). Anonymized data will be saved until 2050. Other researchers may be given access to this material under the approval and supervision of Dr. Rodríguez-González.

Therapists providing therapy as a result of this study will keep client files that contain session notes and relevant case material (e.g., consent to treatment, assessment reports, psychometric test data) under lock and key at their clinics, as per the regulations of the governing bodies of their respective country and the specific region where they have established their private clinical practice. These materials will be destroyed after a 5-year period or once the minimum legal-period set forth by said governing body has been met.

#### Use of video recordings for educational/training purposes

Participating couples will be given the option to allow the video recordings of their therapy sessions to be used for educational/training purposes. Some therapy sessions are particularly useful for showing therapists in training how certain interventions of a specific model are to be carried out. If you agree to the use of your sessions for this purpose:

- The researchers in charge of this study will seek to identify as effective educational material, parts of sessions or entire sessions, in which you participated as a therapy client.
- This educational material will be kept as confidential training material with access requiring a password (secured in the same way as the research data), at the University of Navarra under the responsibility of the primary investigator (IP) and at Brigham Young University under the responsibility of the co-primary investigator (CO-IP).

<sup>&</sup>lt;sup>2</sup> Related legislation in force in each country will be applied.

- This material will be used only in courses taught by members of the research team or by
  members of the departments that are linked to the study, and always under the supervision and
  express consent of the IP of the study, as they are the parties responsible for the custody of
  these materials.
- Additionally, these materials may be used by the therapists and supervisors that directly participate in the study, so long as they are used for educational/training purposes and only in courses in which they are the primary teachers. These therapists and supervisors are not authorized to share or make copies of these materials with/for anyone who is not a part of this study even if they are certified therapists or trainers in the model.

You will be asked about this specific question bellow, in appendix 1, where you will be able to state whether you agree or disagree with this issue.

#### **Data Protection**

Be informed that due to the nature of this study, the data collected through the research process of the study (including your answers to questionnaires and video recordings of your therapy sessions if you are part of the treatment group), will be sent from the country in which they originate to the primary investigators of that study who are at the University of Navarra (in Spain), and in some occasions from there to investigators at Brigham Young University (in the US). These transfers will take place through procedures that will maximize security (a server that will receive the encrypted files securely and which will have a secure login system, which will include dual authentication).

Below we provide legal clauses which explain the handling procedures of your personal information as laid out by the current legislation of the European Union (Regulation 2016/679; Directive 2016/680):

- The party responsible for the handling of your personal information collected in relation to this study is the University of Navarra, Edificio Central, Campus Universitario, Navarra (Spain)
- The study may include the handling of sensitive personal information, for example, information regarding your life and sexual health.
- Data/information from this study may be ceded to Brigham Young University in the United States, which is a country that the European Commission (European Union) has not included in its list of countries which have an equivalent level of data protection to those belonging to the European Union.
- You have the right to remove your consent and to exercise your rights of access, rectification, suppression, opposition, limitation and portability of your personal information at any point in the study.
- You may exercise these rights and pose any questions regarding how your personal information is being handled to the Data Protection Officer at the University of Navarra through the email address <a href="mailto:dpo@unav.es">dpo@unav.es</a>.

You will be asked about this specific question later in appendix 1.

## **QUESTIONS**

Please feel free to ask questions before agreeing to participate. Should you choose to participate, you are encouraged to ask questions throughout and after the research study. Dr. Rodríguez-Gonzalez can be reached at +34 948 425600 Ext. 802367 (Spain phone number), or by email at: effects@unav.es for questions regarding study participation. The Institutional Review Board of Brigham Young University and the University of Navarra have each reviewed this protocol. If you have any questions about your rights as a research participant, you may contact the following Institutional Review Board.

Brigham Young University University of Navarra
Institutional Review Board Institutional Review Board

Phone: 801-422-3841Email: Phone: 948 42 56 00 (Ext. 82 4055)

orca@byu.edu Email: ceic@unav.es

#### **SIGNATURES**

I have read the preceding information and have had a chance to ask questions to help me understand what my participation will involve. My signature below indicates that the research study and related procedures have been explained to me and that I freely give my consent to participate in the research study, unless I decide otherwise (abandon the study). I acknowledge that I will receive a signed copy of this consent form.

| Participant (Print full name) | Signature | Date |
|-------------------------------|-----------|------|

#### RESEARCH ASSISTANT-THERAPIST STATEMENT

I certify that I have explained the research study to the above individual, including the purpose, the procedures, the possible risks and potential benefits associated with participation in this research study. Any questions raised have been answered to the individual's satisfaction. I believe that the participant fully understands my explanations and has freely given informed consent.

| Investigator (Print full name) | Si amatuma | Data |
|--------------------------------|------------|------|
| Investigator (Print full name) | Signature | Date |

## Appendix: Video release

All therapy sessions will be video recorded as is standard therapy practice in many settings. Video recordings will be used for four proposes:

- Supervision [therapists will receive supervision during the study, and they should share video clips with their supervisors to receive feedback on how they can improve their intervention]
- Implementation [once the group treatment end, the video will be used to verify treatment fidelity to the model evaluated; that is, people from the research team will visualize extracts from the sessions to verify that the therapist is performing an Emotionally Focused Therapy intervention, and no other models].
- Research hypothesis [some aspects of the research project need to review the videotaped sessions looking for key-events according to the theoretical model that informs the Emotionally Focused Therapy approach].
- Training [for those couples who accept, some clips of their therapy sessions or a complete session could be used in the future for training proposes to help other therapists learn the model]

| | YES | NO |
|---|---|---|
| I agree with the research uses of the video-tape of my therapy sessions | | |
| (Types of use: supervision, implementation checking, and research hypothesis) | | |
| I agree with the training use of the video-tapes of my therapy sessions but only in | | |
| settings outside my country of residency | | |
| I agree with the training use of the video-tapes of my therapy sessions in settings both | | |
| in my country of residency and in any other country | | |
| Participant (Print full name) Signature Date | | |

As already referred to in the informed consent previously, you should be aware that due to the nature of this study, the data collected through the research process of the study (including your answers to questionnaires and video recordings of your therapy sessions if you are part of the treatment group), will be sent from the country in which they originate to the primary investigators of that study who are at the University of Navarra (in Spain), and in some occasions from there to investigators at Brigham Young University (in the US). This means international transfers that include countries that are not members of the European Union, and therefore are not subject to its legal regulation on the security of personal data protection. These transfers will take place through procedures that will maximize security (a server that will receive the encrypted files through SSL/TLS, and which will have a secure login system, which will include dual authentication). In such circumstances, the transfer will follow applicable Data Protection Law. We take reasonable steps to ensure that the Personal Data is treated securely including using appropriate safeguards such as the Standard Contractual Clauses as approved by the European Commission (European Union).

Withdraw, access and rectification. Pursuant to General Data Protection Regulation (GDPR) you have certain rights to access, transferring or deleting your personal data. Also, you have the right of withdrawing your consent to use your personal videos. For assistance in exercising these rights, please refer to the university data protection webpages or the researchers in charge of the study (you have the contact details in the consent form).

## **SPANISH VERSION**

## Formulario de consentimiento informado para los participantes en el estudio

TÍTULO DEL ESTUDIO DE INVESTIGACIÓN: Terapia de pareja focalizada en las emociones: un ensayo clínico en países de habla hispana.

#### **INVESTIGADORES DEL ESTUDIO:**

Martiño Rodríguez-González, Ph.D.<sup>1</sup>, Shayne Anderson, Ph.D.<sup>2</sup>, Alfonso Osorio, Ph.D.<sup>1</sup>, Paul Greenman, Ph.D.<sup>3</sup>, Marie-France Lafontaine Ph.D.<sup>4</sup>, Patrick Steffen, Ph.D.<sup>2</sup>, Jonathan Sandberg, Ph.D.<sup>2</sup>, María Calatrava, Ph.D.<sup>1</sup>, María del Pilar Martínez-Díaz Ph.D.<sup>5</sup> y estudiantes de posgrado de la UNAV y la BYU. [¹Universidad de Navarra (UNAV), ²Universidad Brigham Young (BYU), ³Universidad de Québec au Outaouais (UQO), ⁴Universidad de Otawa (UO), ⁵Universidad Pontificia de Comillas]

El Dr. Martiño Rodríguez-González (Ph.D.), terapeuta familiar y de pareja, investigador en el Instituto Cultura y Sociedad (ICS) de la Universidad de Navarra, es el investigador principal de este proyecto de investigación. Para cualquier duda, puede ponerse en contacto con él en el edificio de Bibliotecas. E-31009. Universidad de Navarra. Pamplona (España). También por teléfono en: +34 948 425600 Ext. 802367, o por email en: effects@unav.es

| Nombre del participante: |
|--------------------------|
| Fecha: |

#### INTRODUCCIÓN

Se le ha invitado a que participe en un proyecto de investigación. Antes de decidir ser parte de este estudio científico, debe comprender los riesgos y beneficios que puede implicar su participación, para poder tomar una decisión informada. Esto se conoce como consentimiento informado. Este formulario de consentimiento le dará información sobre este proyecto de investigación y lo que implicará participar en él. Si desea obtener más información sobre algo mencionado aquí, o si tiene alguna otra cuestión, no dude en preguntar (Dr. Rodríguez-González, con quien puede contactar por correo postal en: Edificio de Bibliotecas. E-31009. Universidad de Navarra. Pamplona. España. Teléfono al: +34948 425600 Ext. 802367, o por e-mail al effects@unav.es)

Una vez que comprenda lo que implica esta investigación, se le pedirá que firme este formulario de consentimiento si aún desea participar en este estudio. Usted es libre de elegir si desea o no participar. Además, puede abandonar el estudio en cualquier momento, incluso después de que el proyecto de investigación haya comenzado. Si decide abandonar el estudio, como pareja se les reembolsará \$ 100 por cada etapa completada durante su participación (\$50 a cada miembro de la pareja; de esta cantidad será necesario restar los costes en caso de una transacción internacional y/o cambio de divisa). Dado que estamos examinando cómo cambian las parejas durante la terapia, si decide no participar en los elementos del proyecto asociados a la investigación (p. ej., cuestionarios), entonces no se le asignará un terapeuta ni se le proporcionará una terapia complementaria para parejas; sin embargo, si lo desea, sí podemos proporcionarle una lista de servicios comunitarios disponibles en su área.

Antes de firmar este formulario, haga las preguntas que precise sobre cualquier aspecto de este estudio que no le resulte claro. Puede tomarse todo el tiempo que sea necesario para pensar acerca de esta propuesta.

#### **OBJETIVO DEL ESTUDIO**

Esta investigación ha sido diseñada para comprender mejor el impacto que puede tener la terapia en las relaciones de pareja en personas de habla hispana. En otras palabras, el objetivo de este estudio es evaluar si un modelo de terapia en concreto, la terapia focalizada en las emociones, puede ayudar a que las parejas de habla hispana desarrollen una relación más estrecha con su pareja y aprendan cómo mantener esta cercanía una vez la terapia finaliza.

#### **PROCEDIMIENTO**

## ¿Qué implica la participación en este estudio?

Durante esta visita, si decide firmar el formulario de consentimiento y participar en el estudio, se le pedirá que complete una serie de cuestionarios y tenga una entrevista personal con uno de los investigadores/terapeutas del proyecto, para que podamos asegurarnos de que comprende lo que implica participar en el estudio y poder confirmar que cumple los criterios de selección. En estos cuestionarios se le preguntará sobre su personalidad, estado de ánimo, salud y otras cuestiones más generales, así como sobre cómo es su relación de pareja. La entrevista personal durará unos 30-40 minutos (15-20 minutos aproximadamente con cada miembro de la pareja por separado).

Si tras esta primera visita aún sigue siendo un candidato potencial para entrar a formar parte de este estudio, se le notificará por correo electrónico y/o una llamada telefónica en algún momento en los siguientes 2-5 días hábiles posteriores a su visita. Si no cumpliera con los criterios para ser seleccionado, no podrá ser incluido en el estudio. Pero se le proporcionará información sobre clínicas a las que podrá acudir si desea recibir terapia de pareja en la ciudad donde reside. Con independencia de ser elegido o no, sus respuestas se conservarán para poder realizar futuras comparaciones en el estudio, con las respuestas de otros participantes. Sin embargo, sus datos personales serán totalmente eliminados para garantizar el anonimato y la confidencialidad de las respuestas.

Si son seleccionados y deciden participar en el estudio, se les asignará aleatoriamente, junto a su pareja, a uno de estos dos grupos: al "grupo control" o al "grupo tratamiento". Si son asignados al grupo control, se les pedirá que completen una serie de evaluaciones periódicas, así como que participen en una fase de seguimiento con uno o más miembros del equipo de investigación a través de llamadas telefónicas ocasionales durante un período de 5 a 7 meses. Al final de este proceso, se le ofrecerá, junto a su pareja, la oportunidad de participar en un programa psico-educativo para parejas durante un fin de semana. Este programa está basado también en el modelo de la terapia focalizada en las emociones y se llama taller "abrázame fuerte".

Si son asignados al grupo en terapia, se les pedirá que participen en 20 sesiones de terapia de pareja, cada una de estas sesiones tendrá 75 minutos de duración. Generalmente estas sesiones tendrán una frecuencia semanal. Antes y/o después de dichas sesiones de terapia, se les pedirá colaboración para que completen una serie de cuestionarios que forman parte de los elementos del proyecto asociados a la investigación. Todas las sesiones de terapia se realizarán en una clínica de terapia de pareja cercano a su residencia habitual.

Con independencia del grupo al que sea asignado aleatoriamente, completar los cuestionarios después de cada sesión de terapia o en cada punto del proceso de seguimiento, no implicaría más de 10 min. En algunos casos, en lugar de rellenarse en lápiz y papel, se pedirá a los participantes que completen los cuestionarios on-line (en la propia consulta del terapeuta o desde su casa).

## Terapia de pareja

Si forma parte del "grupo tratamiento", se le asignará un terapeuta con experiencia que le llamará para programar su primera cita de terapia junto con su pareja. Recibirán un total de 20 sesiones de terapia con una duración aproximada de 75 minutos cada una. Usted y su pareja deberán asistir a la terapia juntos cada semana. Además, en algún momento entre las sesiones 2 y 5, su terapeuta les recibirá por separado para tener con ustedes una sesión de terapia individual. Todos los terapeutas del estudio están formados en la aplicación de un modelo de terapia llamado Terapia focalizada en las Emociones (TFE). La supervisión del proceso de terapia será realizada por supervisores certificados en este modelo. Todas las sesiones serán grabadas en video y / o grabadas en audio para fines de supervisión y de investigación.

Su decisión de participar en este estudio implica que están dando su aprobación al marco de investigación del mismo. Esto supone aceptar ser grabado en video durante todas las sesiones de terapia y completar los cuestionarios que se le entreguen. Como participante, usted puede decidir abandonar el estudio en cualquier momento. Sin embargo, mientras participe en él, asume explícitamente estar haciéndolo consciente de la naturaleza del estudio.

#### Modelo terapéutico utilizado en este estudio de investigación

El modelo específico de la terapia de pareja que se le ofrecerá se llama terapia de pareja focalizada en las emociones (TFE). La terapia de pareja focalizada en las emociones considera que los conflictos en una relación son resultado de ciclos negativos de interacción que las parejas desarrollan con el tiempo. La TFE ayuda a los miembros de la pareja a salir de estos patrones negativos de comportamiento, para que puedan ayudarse mutuamente a establecer seguridad y conexión dentro de su relación. También les enseña cómo solicitar y responder mejor a las necesidades de apoyo y amor del otro. Los estudios científicos han demostrado de modo consistente que este modelo de terapia es muy útil para ayudar a las parejas con dificultades a mejorar su relación, y que estas mejoras permanezcan en el tiempo, incluso una vez finalizada la terapia.

## ¿Cuánto me costará participar? ¿Me pagarán por participar?

La participación en el estudio <u>no</u> conlleva ningún gasto asociado. Al contrario, cada pareja recibirá \$60.00 por cada hora dedicada a colaborar con los aspectos de investigación (p. ej., completar cuestionarios; esto excluye el tiempo dedicado a la asistencia a las sesiones de terapia). Calculamos que esta dedicación puede suponer un tiempo de 7 horas durante los meses que dura el estudio, en función del grupo al que sean asignados. Se les pagará \$80 (por pareja) por cada hora adicional a las 7 horas estimadas.

A las parejas asignadas al grupo de tratamiento se les pedirá que participen en una fase de seguimiento una vez que se hayan completado las intervenciones terapéuticas (las 20 sesiones de terapia). Este seguimiento no se solicitará a las parejas que hayan estado en el grupo control y vayan a participar en la intervención de tipo psicoeducativo basada en el modelo de la TFE (llamada "abrázame fuerte"). Las evaluaciones de seguimiento se realizarán a los 3, 6, 12, 18 y 24 meses después de que se hayan completado las 20 sesiones de terapia. Las parejas que completen las dos primeras evaluaciones de seguimiento, que tendrán lugar a los 3 y a los 6 meses, recibirán \$ 70 (por pareja). De manera adicional, recibirán \$ 70 por completar la evaluación a los 12 y a los 18 meses. Finalmente, recibirán \$ 70 más por completar la evaluación a los 24 meses de haber finalizado la terapia.

#### **RIESGOS Y BENEFICIOS**

<u>Riesgos:</u> Su participación en la terapia implicará que tenga que responder a preguntas sobre sus propios pensamientos y emociones, además de completar los cuestionarios del estudio. Los participantes pueden

experimentar alguna molestia al responder, parecida a si recordaran un evento triste en sus vidas. Si por alguna razón esto sucediera y las molestias fueran difíciles de manejar por parte de los participantes, se les sugerirá que hablen de ello con su terapeuta, por ser un profesional de la salud mental cualificado. Los participantes pertenecientes al grupo de control recibirán la información de contacto del Dr. Martiño Rodríguez-González, un psicólogo registrado, en caso de que deseen abordar cualquier molestia que pueda surgir.

<u>Beneficios</u>: Los beneficios de participar en un proceso de terapia siguiendo el modelo de la TFE están bien establecidos. Estos incluyen la mejora en la relación de pareja, así como en el estado de ánimo y el estado psicológico general.

#### **CONFIDENCIALIDAD**

Toda la información recogida durante el estudio será tratada con la máxima confidencialidad y todos los datos personales serán protegidos. Los cuestionarios que usted complete, las notas de su psicoterapeuta y los registros de audio y/o video utilizados en este estudio se guardarán en un archivador cerrado con llave en la clínica de psicoterapia o el lugar donde se llevan a cabo sus sesiones de terapia. Todos los cuestionarios on-line se completarán y almacenarán en un servidor seguro y encriptado. Además, esta información se enviará a la Universidad de Navarra a través de un canal de comunicaciones seguro y codificado. No se escribirán nombres ni información personal que vincule su identidad y la de su pareja con sus respuestas a los cuestionarios o a los registros de video, sino que se enlazarán a través de algún código interno. Sus nombres solo serán conocidos por el personal que participa directamente en el estudio de investigación. Estos incluyen a los investigadores del estudio, los supervisores clínicos y su terapeuta. Por último, queda garantizado el anonimato en las publicaciones científicas que se deriven de sus datos de modo que ningún individuo o pareja podrá ser identificado.

Sin embargo, si se dan algunas situaciones, un miembro del equipo de investigación debe romper este acuerdo de confidencialidad<sup>3</sup>. Estas situaciones son excepcionales y hacen referencia a casos en los que haya una orden judicial, casos de peligro inminente para usted o para otros, casos en los que haya un conocimiento de abuso infantil u otro tipo de abusos por parte de un profesional de la salud. En cuanto al abuso infantil, la ley exige a los investigadores que informen a las autoridades correspondientes si tienen conocimiento de que un niño menor de 18 años está siendo abusado o en riesgo de ser abusado. Esto es diferente a que usted pudiera manifestar haber sido víctima de abuso infantil. Solo si revelara que existe la posibilidad de que su abusador pudiera estar en contacto con niños en ausencia de supervisión, será necesario poner en conocimiento de las autoridades correspondientes.

## Almacenamiento de datos para fines de investigación

Una copia digital de los cuestionarios de papel y lápiz (que va a responder en la consulta de su terapeuta) y de la lista que vincula su nombre y el de su pareja con un código anónimo de identificación, así como otra información de contacto (por ejemplo, el correo electrónico), se guardará en un disco duro con contraseña en un archivador cerrado con llave en el despacho del Dr. Rodríguez-González por un período de 5 años una vez finalizado el estudio, transcurrido lo cual esa información será destruida. Solo el investigador principal, el Dr. Rodríguez-González, tendrá acceso a esta información.

Todos los demás archivos impresos y electrónicos (no mencionados en el párrafo previo) relacionados con este proyecto de investigación (por ejemplo, matriz de datos con los cuestionarios codificados o sesiones de terapia grabadas en video) se guardarán en un disco duro con contraseña en un archivador cerrado con llave en la oficina del Dr. Rodríguez-González (UNAV) por un período de 15 años

<sup>&</sup>lt;sup>3</sup> Se aplicará la legislación relacionada vigente en cada país.

(2035). Los datos anónimos se guardarán hasta 2050. Otros investigadores podrán tener acceso a este material anónimo bajo la aprobación y supervisión del Dr. Rodríguez-González.

Los terapeutas que ofrecen terapia en el marco de este estudio conservarán los archivos de los clientes que contienen notas de la sesión y material relevante del caso (p. ej., consentimiento para la terapia, informes de evaluación, datos de los cuestionarios) bajo llave en sus clínicas, de acuerdo con las regulaciones del gobierno y organismos de sus respectivos países y la región específica donde han establecido su práctica clínica privada. Estos materiales serán destruidos totalmente después de un período de 5 años o una vez que se haya cumplido el período legal mínimo establecido por dicho órgano rector de su país de ejercicio profesional.

## Uso de las grabaciones en video para fines de entrenamiento o formación

Las parejas participantes tendrán la opción de permitir que las grabaciones de video de sus sesiones de terapia se utilicen con fines educativos y/o formativos. Algunas sesiones de terapia son particularmente útiles para mostrar a los terapeutas en procesos de formación cómo se deben realizar ciertas intervenciones de un modelo específico. Si acepta el uso de sus sesiones para este propósito:

- Los investigadores a cargo de este estudio buscarán identificar como material educativo efectivo, partes de sesiones o sesiones enteras, en las que participó como cliente de terapia.
- Este material educativo se mantendrá como material confidencial con acceso a través de contraseña (protegida de la misma manera que los datos de la investigación), en la Universidad de Navarra bajo la responsabilidad del investigador principal (IP) y en la *Brigham Young University* bajo la responsabilidad del co-investigador principal (CO-IP).
- Este material se usará solo en cursos impartidos por miembros del equipo de investigación o por otras personas vinculadas directamente al estudio, y siempre bajo la supervisión y el consentimiento expreso del investigador principal del estudio, ya que es el responsable de la custodia de estos materiales.
- Además, estos materiales audiovisuales pueden ser utilizados por los terapeutas y supervisores que participan directamente en el estudio, siempre que se utilicen con fines educativos o/ formativos, y solo en los cursos en los que ellos mismos son los entrenadores o ponentes principales. Estos terapeutas y supervisores no están autorizados para compartir con o hacer copias de estos materiales con otras personas que no hayan participado en el estudio, aunque estos sean terapeutas o entrenadores certificados en el modelo.

Se le preguntará más adelante por esta cuestión específica, en el apéndice 1, donde puede manifestar si está de acuerdo o no con este uso.

#### Protección de datos

Tenga en cuenta que, debido a la naturaleza de este estudio, los datos recopilados a través del proceso de investigación del estudio (incluidas sus respuestas a cuestionarios y grabaciones de video de sus sesiones de terapia si es parte del grupo de tratamiento), se enviarán desde el país en el que se originan a los investigadores principales de ese estudio que están en la Universidad de Navarra (en España), y en algunas ocasiones a investigadores de la Brigham Young University (en los Estados Unidos). Estas transferencias se llevarán a cabo mediante procedimientos que maximizarán la seguridad (un servidor que recibirá los archivos cifrados de forma segura y que tendrá un sistema de inicio de sesión seguro, que incluirá autenticación dual).

A continuación, le ofrecemos las cláusulas legales que explican los procesos de tratamiento de su información personal de acuerdo a lo que establece la legislación vigente de la Unión Europea (Regulation 2016/679; Directive 2016/680):

- La entidad responsable del tratamiento de su información personal recopilada en relación con este estudio es la Universidad de Navarra, Edificio Central, Campus Universitario, Navarra (España)
- Este estudio puede incluir el manejo de información personal sensible, como por ejemplo, información sobre su vida y salud sexual.
- Los datos / información de este estudio pueden ser cedidos a la Brigham Young University en los Estados Unidos, que es un país que la Comisión Europea (Unión Europea) no ha incluido en su lista de países que tienen un nivel equivalente de protección de datos a los que pertenecen a la Unión Europea.
- Tiene derecho a retirar su consentimiento y a ejercer sus derechos de acceso, rectificación, supresión, oposición, limitación y portabilidad de su información personal en cualquier momento del estudio.
- Puede ejercer estos derechos y plantear cualquier pregunta sobre cómo se maneja su información personal a la Oficina de Protección de Datos de la Universidad de Navarra a través de la dirección de correo electrónico dpo@unav.es.

Se le preguntará más adelante por esta cuestión específica, en el apéndice 1.

#### **PREGUNTAS**

No dude en hacer las preguntas que necesite antes de aceptar participar. Si decide participar, se le anima a que haga preguntas las preguntas que desee también durante y después del estudio de investigación. Puede ponerse en contacto con el Dr. Rodríguez-González a través del teléfono +34948 425600 Ext. 802367 (número de teléfono de España), o por correo electrónico a: effects@unav.es para preguntas relacionadas con su participación en el estudio. Los comités de ética de la Brigham Young University y de la Universidad de Navarra han revisado este protocolo. Si tiene alguna pregunta sobre sus derechos como participante en la investigación, puede comunicarse con los comités de ética de estas universidades:

Universidad de Navarra **Brigham Young University** Institutional Review Board Comité de ética de la investigación Phone: 948 42 56 00 (Ext. 82 4055) Phone: 801-422-3841 Email: ceic@unav.es Email: orca@byu.edu

#### **FIRMAS**

Participante (escriba nombre y apellidos)

He leído la información recogida en este documento y he tenido la oportunidad de hacer preguntas para ayudarme a comprender en qué consistirá mi participación. Mi firma a continuación indica que se me ha explicado claramente el estudio y los procedimientos relacionados con el mismo, y que doy libremente mi consentimiento para participar en esta investigación, mientras no decida lo contrario (abandonar el estudio). Tengo conocimiento de que recibiré una copia firmada de este formulario de consentimiento.

| ransopanie (eserieu nemero y upomues) | | 1 001100 |
|---|---|---|
| <b>DECLARACIÓN DEL ASISTENTE DE INVESTI</b> Certifico que le he explicado el proyecto de investigad incluidos los objetivos, procedimientos, posibles participación en este estudio. Cualquier pregunta plante el participante comprende completamente mis expliinformado. | ción a la persona res<br>riesgos y posibles<br>eada ha sido satisfac | gistrada previamente en el texto,<br>beneficios asociados con su<br>toriamente respondida. Creo que |
| Investigador/terapeuta (escriba nombre y apellidos) | Firma | Fecha |

Firma

Fecha

su

#### Apéndice: Difusión en video

Todas las sesiones de terapia se grabarán en video como es habitual en la práctica terapéutica en muchos modelos. Las grabaciones de video se utilizarán para cuatro fines:

- Supervisión [los terapeutas recibirán supervisión durante el estudio, y deberán compartir cortes de video de las sesiones de terapia con sus supervisores para recibir comentarios sobre cómo pueden mejorar su intervención]
- Implementación [una vez que finalice el tratamiento, el video se utilizará para verificar la fidelidad al modelo
  que se quiere evaluar; es decir, personas del equipo de investigación visualizarán extractos de las sesiones
  para comprobar que el terapeuta está realizando una intervención desde la terapia focalizada en las
  emociones, y no otros modelos].
- Hipótesis de investigación [algunos aspectos del proyecto de investigación necesitan revisar las sesiones grabadas en video buscando eventos clave de acuerdo con el modelo teórico que informa el enfoque centrado emocionalmente].
- Formación/docencia [opcionalmente, solo para aquellas parejas que lo decidan, algunos cortes de vídeo de sus sesiones de terapia o alguna sesión completa podrían usarse en el futuro para fines docentes (p. ej., la formación de nuevos terapeutas que están aprendiendo el modelo)]

| | SÌ | NO |
|---|---|---|
| Estoy de acuerdo con el uso de mis videos de las sesiones de terapia para fines de | | |
| investigación (lo que incluye los fines: supervisión, implementación e hipótesis de investigación) | | |
| Estoy de acuerdo con el uso de las grabaciones de mis sesiones de terapia para fines | | |
| docentes, pero solo en entornos fuera de mi país de residencia | | |
| Estoy de acuerdo con el uso de las grabaciones de mis sesiones de terapia para fines | | |
| docentes, tanto en mi país de residencia como fuera de él | | |

| Participante (escriba nombre y apellidos) | Firma | Fecha |
|-------------------------------------------|-------|-------|

Como ya fue referido en el consentimiento informado previamente, usted debe tener en cuenta que los datos recopilados a través del proceso de investigación (incluidas sus respuestas a cuestionarios y grabaciones de video de sus sesiones de terapia si es parte del grupo de tratamiento), se enviarán desde el país en el que se originan a los investigadores principales de ese estudio que están en la Universidad de Navarra (en España), y en algunas ocasiones a investigadores de la *Brigham Young University* (en los Estados Unidos). Esto significa transferencias internacionales que incluyen a países que no son miembros de la Unión Europea, y por tanto no están sujetos a su regulación legal en materia de seguridad de protección de datos personales. Estas transferencias de datos se llevarán a cabo mediante procedimientos que maximizarán la seguridad (un servidor que recibirá los archivos cifrados a través de SSL / TLS, y que tendrá un sistema de inicio de sesión seguro, que incluirá autenticación dual). En dichas circunstancias, la transferencia de datos seguirá la Ley de Protección de Datos aplicable. Tomaremos las medidas oportunas para garantizar que los datos personales se traten de forma segura, incluyendo las garantías asociadas a la normativa de protección de datos estándar aprobada por la Comisión Europea (Unión Europea).

| He entendido todas las condiciones del estudio y quiero participar en él. Estoy de | | N. ( ) |
|---|---|---|
| acuerdo con la transferencia internacional de las grabaciones de video de las sesiones | Si ( ) | No ( ) |
| de terapia y de otros documentos que puedan ser necesarios vinculados con el estudio | | |

Retirada, acceso y rectificación. De conformidad con el Reglamento General de Protección de Datos (GDPR), usted tiene ciertos derechos para acceder, transferir o eliminar sus datos personales. Además, tiene derecho a retirar su consentimiento para usar sus videos personales. Para obtener ayuda en el ejercicio de estos derechos, consulte las páginas web de protección de datos de la universidad o de los investigadores a cargo del estudio (tiene los datos de contacto en el formulario de consentimiento.